CLINICAL TRIAL: NCT00908583
Title: Desensitization for Preformed Anti-HLA Antibodies in Kidney Transplantation
Brief Title: Desensitization in Kidney Transplantation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, E. Steve Woodle, MD, FACP, University of Cincinnati
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: X05295
Record Dates: First submitted 2009-05-26; First posted 2009-05-27 (Estimated); Results first posted 2016-02-26 (Estimated); Last update posted 2016-04-01 (Estimated); Status verified 2016-03

CONDITIONS: HLA Sensitization
Keywords: Alloantibody; Desensitization; Kidney Transplantation; Nephrology; Plasma Cells; Translational Research/Science
MeSH Terms: interventions — Plasmapheresis; Bortezomib; Rituximab; Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Phase 1, two stages (Experimental): Patients will receive 1 dose of rituximab, 4 doses of bortezomib and plasmapheresis. Rituximab will be given at a dose of 375 mg/m2 on day 32. Patients will receive 1.3 mg/m2 of bortezomib via intravenous push (IVP) over 3-5 seconds. Bortezomib will be administered on days 1, 4, 8, and 11. For those patients who go on to Stage 2 of desensitization, bortezomib will be administered via IV push over 3-5 seconds during the pre-transplant period on days 32, 35, 39, 42. Methylprednisolone will be administered within 30 minutes of each bortezomib administration in both stages of desensitization. With the first and second doses, administer methylprednisolone 100mg via IV push. With the third and fourth doses, administer methylprednisolone 50mg IVP.
  Interventions: Drug: plasmapheresis; Drug: Bortezomib; Drug: Rituximab; Drug: Methylprednisolone
- Phase 2, two stages (Experimental): Patients will receive 1 dose of rituximab, 4 doses of bortezomib and plasmapheresis. Rituximab will be given at a dose of 375 mg/m2 on day -7. Patients will receive 1.3 mg/m2 of bortezomib via intravenous push (IVP) over 3-5 seconds. Bortezomib will be administered on days 1, 4, 8, and 11. For those patients who go on to Stage 2 of desensitization, bortezomib will be administered via IV push over 3-5 seconds during the pre-transplant period on days 32, 35, 39, 42. Methylprednisolone will be administered within 30 minutes of each bortezomib administration in both stages of desensitization. With the first and second doses, administer methylprednisolone 100mg via IV push. With the third and fourth doses, administer methylprednisolone 50mg IVP.
  Interventions: Drug: plasmapheresis; Drug: Bortezomib; Drug: Rituximab; Drug: Methylprednisolone
- Phase 3, two stages (Experimental): Patients will receive 1 dose of rituximab and 4 doses of bortezomib. Rituximab will be given at a dose of 375 mg/m2 on day -7. Patients will receive 1.3 mg/m2 of bortezomib via intravenous push (IVP) over 3-5 seconds. Bortezomib will be administered on days 1, 4, 8, and 11. For those patients who go on to Stage 2 of desensitization, bortezomib will be administered via IV push over 3-5 seconds during the pre-transplant period on days 23, 26, 30 and 33. Methylprednisolone will be administered within 30 minutes of each bortezomib administration in both stages of desensitization. With the first and second doses, administer methylprednisolone 100mg via IV push. With the third and fourth doses, administer methylprednisolone 50mg IVP.
  Interventions: Drug: plasmapheresis; Drug: Bortezomib; Drug: Rituximab; Drug: Methylprednisolone
- Phase 4, single stage (Experimental): Patients will receive 1 dose of rituximab and 6 doses of bortezomib. Rituximab will be given at a dose of 375 mg/m2 on day -7. Patients will receive 1.3 mg/m2 of bortezomib via intravenous push (IVP) over 3-5 seconds. Bortezomib will be administered during the pre-transplant period on days 1, 4, 8, and 11, 14, and 17. Methylprednisolone will be administered within 30 minutes of each bortezomib administration in both stages of desensitization. With the first and second doses, administer methylprednisolone 100mg via IV push. With the third and fourth doses, administer methylprednisolone 50mg IVP.
  Interventions: Drug: plasmapheresis; Drug: Bortezomib; Drug: Rituximab; Drug: Methylprednisolone
- Phase 5, single stage (Experimental): Phase 5 evaluated even greater bortezomib dosing density by eliminating the inter-cycle dosing interval. Phase 5 evaluated eight consecutive doses of bortezomib with one dose of rituximab. Rituximab will be given at a dose of 375 mg/m2 on day -7. Patient will receive 1.3 mg/m2 of bortezomib via intravenous push (IVP) over 3-5 seconds. Bortezomib will be administered on days 1, 4, 8, 11, 14, 17, 20, and 23. Methylprednisolone will be administered within 30 minutes of each bortezomib administration in both stages of desensitization. With the first and second doses, administer methylprednisolone 100mg via IV push. With the third and fourth doses, administer methylprednisolone 50mg IVP.
  Interventions: Drug: plasmapheresis; Drug: Bortezomib; Drug: Rituximab; Drug: Methylprednisolone

INTERVENTIONS:
Drug: plasmapheresis — Patients will receive plasmapheresis 1.5 x plasma volume prior to each Bortezomib dose. Plasma volume replacement will be per physician discretion.
Drug: Bortezomib — Patients will receive bortezomib as described in protocol
  Other Names: Velcade
Drug: Rituximab — Patients will receive rituximab as described in protocol
  Other Names: Rituxan
Drug: Methylprednisolone — Each bortezomib dose will be preceded by intravenous methylprednisolone (100mg for first two doses and 50mg for following doses).
  Other Names: Medrol

SUMMARY:
To determine if deletional strategies will provide effective desensitization.

DETAILED DESCRIPTION:
A prospective iterative trial of proteasome inhibitor (PI)-based therapy for reducing HLAantibody (Ab) levels was conducted in five phases differing in bortezomib dosing density and plasmapheresis timing. Phases included 1 or 2 bortezomib cycles (1.3mg/m2,6-8 doses), one rituximab dose and plasmapheresis. HLA Abs were measured by solid phase and flow cytometry (FCM) assays. Immunodominant Ab (iAb) was defined as highest HLA Ab level. Forty-four patients received 52 desensitization courses (7 patients enrolled in multiple phases): Phase 1 (n=20), Phase 2 (n=12), Phase 3 (n=10), Phase 4 (n=5), Phase 5 (n=5).

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65
* Voluntary written informed consent
* Patient on deceased donor wait list with a current or peak cytotoxic or calculated panel reactive antibody (PRA) > 20%

Exclusion Criteria:

* Myocardial infarction within 6 months
* Patient received investigational drug within 14 days prior to initiation of study treatment
* Serious medical or psychological illness
* Diagnosed with malignancy within three years, except complete research of basal cell carcinoma or squamous cell carcinoma of skin, an insitu malignancy or low risk prostate cancer after curative therapy
* Absolute neutrophil count (ANC) < 1000
* Receipt of live vaccine within 4 weeks of study entry
* Female subject that is breast feeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2009-05; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: E. Steve Woodle, MD, Principal Investigator — University of Cincinnati
Locations (2):
- United States (2):
  - The Christ Hospital, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects could be enrolled in multiple study phases. Enrollment in phases 1-2 was an adaptive approach and was fixed a priori in Phases 3-5. The adaptive approach was based on treatment effect (immunodominant antibody (iAb) reduction).
Pre-assignment Details: 44 subjects received 52 treatments in this study. 7 subjects were enrolled in multiple phases. Four patients received treatment in two study phases (two patients were enrolled in Phases 1 and 2, one patient was enrolled in study Phases 1 and 3, and one patient was enrolled in Phases 2 and 3). One patient was enrolled in Phases 1, 2 and 4.
Groups:
- All Study Participants: Combined study participants all phases.
Period: Phase 1
Arm/Group | All Study Participants
Started | 20
Completed | 15
Not Completed | 5
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 4
Period: Phase 2
Arm/Group | All Study Participants
Started | 12
Completed | 10
Not Completed | 2
Not completed — Physician Decision | 1
Not completed — Adverse Event | 1
Period: Phase 3
Arm/Group | All Study Participants
Started | 10
Completed | 8
Not Completed | 2
Not completed — Adverse Event | 2
Period: Phase 4
Arm/Group | All Study Participants
Started | 5
Completed | 3
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Physician Decision | 1
Period: Phase 5
Arm/Group | All Study Participants
Started | 5
Completed | 2
Not Completed | 3
Not completed — Adverse Event | 3

BASELINE CHARACTERISTICS:
Population: Forty-four patients received 52 desensitization courses (7 patients enrolled in multiple phases): Phase 1 (n=20), Phase 2 (n=12), Phase 3 (n=10), Phase 4 (n=5), Phase 5 (n=5). "n" refers to the number of patients. Since patients were enrolled in multiple phases the numbers reported show the total enrollment of each phase.
Groups:
- All Study Participants: Combined study participants, all phases.
Arm/Group | All Study Participants
Number analyzed (Participants) | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.2 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 16
  White | 28
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 44

OUTCOME MEASURES:

1. Secondary Outcome: Overall Safety of Bortezomib
Description: Incidence of grade 3 and above non-hematologic toxicities. Incidence of grade 4 hematologic toxicities. Incidence of all grades of peripheral neuropathy. Incidence of Cytomegalovirus (CMV), Polyomavirus Allograft Nephropathy (PVN), and Posttransplant Lymphoproliferative Disorder (PTLD).
Time Frame: Study Day 62
Measure: Number; unit: participants
Groups:
- Phase 1, Cycle 1; Phase 1 Cycle 2; Phase 2, Cycle 1; Phase 2 Cycle 2; Phase 3, Cycle 1; Phase 3, Cycle 2: Deletional, two stage approach with terminal plasmapheresis
  Deletional therapy/plasmapheresis: B lymphocyte/plasma cell deletional therapy will be administered
- Phase 4, Single Stage: Deletional, one stage approach with six doses of plasmapheresis prior to each bortezomib dose
  Deletional therapy/plasmapheresis: B lymphocyte/plasma cell deletional therapy will be administered
- Phase 5, Single Stage: Deletional, one stage approach with eight doses of plasmapheresis prior to each bortezomib dose
  Deletional therapy/plasmapheresis: B lymphocyte/plasma cell deletional therapy will be administered
Arm/Group | Phase 1, Cycle 1 | Phase 1 Cycle 2 | Phase 2, Cycle 1 | Phase 2 Cycle 2 | Phase 3, Cycle 1 | Phase 3, Cycle 2 | Phase 4, Single Stage | Phase 5, Single Stage
Number analyzed (Participants) | 19 | 16 | 11 | 10 | 10 | 8 | 4 | 5
participants
  Incidence of CTCAE Grade 3 Anemia (<8.0-6.5 g/dL) | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 1
  Incidence of CTCAE Grade 4 Anemia (<6.5g/dL) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Incidence of CTCAE Grade 3 Thrombocytopenia | 1 | 2 | 0 | 0 | 1 | 1 | 0 | 0
  Incidence of CTCAE Grade 4 Thrombocytopenia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Incidence of CTCAE Grade 3 Neutropenia | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Incidence of CTCAE Grade 4 Neutropenia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Incidence of new onset level 1 PN | 1 | 0 | 3 | 2 | 0 | 1 | 0 | 1
  Incidence of new onset level 2 PN | 5 | 3 | 2 | 3 | 2 | 1 | 0 | 0
  Incidence of new onset level 3 PN | 1 | 3 | 0 | 0 | 1 | 0 | 0 | 0
  Incidence of new onset level 4 PN | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
  Incidence of new onset level 5 PN | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  CMV D+/R- Status | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CMV Viremia or Invasive Disease | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Polyomavirus Allograft Nephropathy (PVN) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Malignancy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Living Donor Transplant Candidates That Are Transplanted
Description: Number of living donor transplant candidates who convert to a negative flow T- and B-cell crossmatch via desensitization and are subsequently transplanted
Time Frame: 1 year post baseline
Measure: Number; unit: participants
Groups:
- All Study Participants: All study participants combined. Counting participants only once even though 7 participants were enrolled in multiple phases.
Arm/Group | All Study Participants
Number analyzed (Participants) | 44
participants | 19

3. Secondary Outcome: Number of Patients Whose Cytotoxic Panel Reactive Antibody (PRA) is Decreased by 50%
Description: Number of patients on the waiting list whose cytotoxic PRA is decreased by 50%.
Time Frame: 46 days
Measure: Number; unit: participants
Groups:
- All Study Participants: All study participants combined.4 participants were enrolled in multiple groups or phases. They are only counted once.
Arm/Group | All Study Participants
Number analyzed (Participants) | 44
participants | 6

4. Secondary Outcome: Acute Rejection Rate
Description: Acute rejection rate at 6 months of all desensitized and transplanted patients
Time Frame: 6 months post transplant
Population: One graft loss occurred due to graft thrombosis within 24 hours (due to unrecognized hypercoagulability disorder without AMR). Two patients were transplanted at other centers and data was not available. This dropped the number of analyzed patients to 16 from 19.
Measure: Number; unit: participants
Groups:
- All Transplanted Participants: Combined phases, transplanted patients.
Arm/Group | All Transplanted Participants
Number analyzed (Participants) | 16
participants | 3

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Phase 1, Two Stages; Phase 2, Two Stages; Phase 3: Deletional, two stage approach with terminal plasmapheresis
  Deletional therapy/plasmapheresis: B lymphocyte/plasma cell deletional therapy will be administered
Arm/Group | Phase 1, Two Stages | Phase 2, Two Stages | Phase 3 | Phase 4, Single Stage | Phase 5, Single Stage
Serious Adverse Events (participants affected / at risk) | 6/20 | 1/12 | 4/10 | 2/5 | 2/5
Other Adverse Events (participants affected / at risk) | 2/20 | 4/12 | 4/10 | 0/5 | 1/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1, Two Stages (N=20) | Phase 2, Two Stages (N=12) | Phase 3 (N=10) | Phase 4, Single Stage (N=5) | Phase 5, Single Stage (N=5)
Generalized Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Patient admitted to hospital 6 days after completing the first bortezomib cycle for generalized weakness and malaise, which subsequently spontaneously resolved.
Pancreatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Patient admitted to the hospital with upper abdominal pain and slight elevation in lipase, but with normal amylase. Pain resolved within 48 hours and lipase returned to normal and was discharged. Event occurred during bortezomib therapy.
Elevated Liver Function Test (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Eight days after the last bortezomib dose of cycle 1, patient developed malaise, nausea, vomiting. Evaluation revealed elevated liver enzymes (aspartate aminotransferase (AST) and alanine aminotransferase (ALT) which both spontaneously resolved.
Chest Pain (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Patient developed chest pain at home with radiation to his left shoulder. Patient has a history of similar chest pain episodes. EKG was normal and troponins negative and patient was discharged from the hospital.
Seizure (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea/Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypoxemia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral Neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Patient experienced atrial fibrillation during routine dialysis at his local dialysis center. Patient was transferred to a local ER where elective cardioversion was performed. The patient fully recovered in the ER.
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blurred Vision (Eye disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Perivascular Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Facial Weakness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1, Two Stages (N=20) | Phase 2, Two Stages (N=12) | Phase 3 (N=10) | Phase 4, Single Stage (N=5) | Phase 5, Single Stage (N=5)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Upper Respiratory Infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Peripheral Sensory Neuropathy (PN) (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper Respiratory Viral Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiopulomonary Instability (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No